CLINICAL TRIAL: NCT06838793
Title: Quality of Recovery After Video-assisted Thoracoscopic Surgery: A Prospective, Randomised, Double-Blinded Trial Comparing Single and Three Level Intertransverse Process Block.
Brief Title: ITPB 1 vs 3 in VATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025.547
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Intertransverse Process Block; Video-assisted Thoracscopic Surgery; Quality of Recovery
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Level Intertransverse Process Block (Active Comparator): Patients with primary carcinoma lung scheduled for resection under VATS procedure and randomized in SL group will receive a single level ITPB at retro SCTL space injection and it will be performed at T5 vertebral level after which two subsequent IM sham injections with 2-3 ml 0.9% saline will be performed at T3 and T7 level.
  Interventions: Procedure: Single Level Intertransverse Process Block
- Three Level Intertransverse Process Block (Active Comparator): Patients with primary carcinoma lung scheduled for resection under VATS procedure and randomized in TL group will receive injection at T3, T5 and T7.
  Interventions: Procedure: Three Level Intertransverse Process Block

INTERVENTIONS:
Procedure: Single Level Intertransverse Process Block — Patients will then be positioned in the lateral decubitus position with the side to be blocked facing upwards, the neck slightly flexed and the upper arm resting on the pillow for the USG ITPB.
  The thoracic intervertebral levels (T3, T5, T7) will be identified and marked on the patient. Ultrasound gel will be applied to the skin foracoustic coupling and the transducer is placed 2-3 cm lateral to the spinous process, at the target vertebral level, in the t After obtaining the target transverse ultrasound window at the articular process level, under strict aseptic precautions and local infiltration (Lignocaine 1%), a SonoTap nerve block needle (Pajunk, 22G, 80 mm, Pajunk, Geisingen, Germany) will be inserted in-plane and slowly advanced from a lateral to medial direction until its tip is located at the medial aspect of the retro-SCTL space. After negative heme aspiration, 25 ml of LA mixture containing 0.5% ropivacaine with 1: 200,000 adrenaline will be injected slowly in small aliquots.
  Arms: Single Level Intertransverse Process Block
Procedure: Three Level Intertransverse Process Block — Patients will then be positioned in the lateral decubitus position with the side to be blocked facing upwards, the neck slightly flexed and the upper arm resting on the pillow for the USG ITPB. After obtaining the target transverse ultrasound window at the inferior articular process level (described above) at the T7 level, under strict aseptic precautions and local infiltration (Lignocaine 1%), a SonoTap nerve block needle (Pajunk, 22G, 80 mm, Pajunk, Geisingen, Germany) will be inserted in-plane and slowly advanced from a lateral to medial direction until its tip is located at the medial aspect of the retro-SCTL space. After negative heme aspiration, 8 ml of LA mixture containing 0.5% ropivacaine with 1:200,000 adrenaline will be injected slowly in small aliquots. Subsequently, similar injections will be performed at T5 and T3 level with 8 ml and 9 ml LA mixture, respectively (Total LA mixture volume: 25 ml).
  Arms: Three Level Intertransverse Process Block

SUMMARY:
This study aims to evaluate the quality of recovery after video-assisted thoracoscopic surgery (VATS) by comparing the efficacy of a single-level intertransverse process block (ITPB) against a three-level ITPB, with particular attention to the quality of recovery measured by the QoR15 score at 24 hours post-surgery.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgeries (VATS) are currently the preferred technique for treating carcinoma lung. Despite being minimally invasive, VATS is associated with significant acute and chronic postoperative pain. Regional anesthetic techniques have the potential to block afferent nociception at the peripheral nerve level, the dorsal root ganglion (DRG), the thoracic sympathetic ganglion, or through a combination of these mechanisms. While the peripheral nerve block techniques such as the intercostal nerve block and serratus anterior plane block can provide analgesia for port related somatic pain, the visceral pain mediated via the thoracic sympathetic chain during VATS procedure are amenable only to epidural or paravertebral regional anaesthetic techniques. The thoracic paravertebral block (TPVB) provides ipsilateral, segmental, somatic, and sympathetic nerve blockade across multiple contiguous thoracic dermatomes and is currently the first choice for VATS. During a TPVB, the local anaesthetic (LA) is injected into the paravertebral space adjacent to the thoracic vertebra, near the intervertebral foramen.

Traditionally, TPVB is performed using either landmark or ultrasound guidance, with the LA deposited anterior to the superior costotransverse ligament (SCTL). This typically involves the block needle piercing the SCTL to reach the wedge-shaped TPVB space. While Thoracic Paravertebral Block (TPVB) is generally regarded as safe, the proximity of the needle tip to the pleura during injection poses a heightened risk of pleural puncture and pneumothorax, especially when administered by less experienced physicians. Consequently, the Erector Spinae Plane Block (ESPB) is gaining popularity as an alternative. However, it is important to note that ESPB also has its own limitations.

Recent advancements have redefined thoracic paravertebral anatomy, identifying a fat-filled retro-SCTL space located behind the SCTL. This space is farther from the pleura but remains in close proximity to anterior neural targets such as the thoracic spinal nerve, the DRG and thoracic sympathetic ganglion. It is hypothesised that an LA injection into the retro-SCTL space-referred to as the Intertransverse Process Block (ITPB) at the medial retro SCTL space-could produce a rapid onset of ipsilateral and/or bilateral segmental somatic and sympathetic nerve blockade of the thoracic dermatomes without the need to pierce the SCTL, thereby reducing the risk of pleural puncture and pneumothorax. Preliminary investigations on the ITPB for VATS is promising, however, there is a paucity of data on the effect of the number of injections following an ultrasound-guided (USG) ITPB on the analgesic efficacy, which this study aims to evaluate.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* 18 to 80 years of age
* Patients with primary carcinoma lung scheduled for resection under VATS procedure

Exclusion Criteria:

* Patient refusal
* Local skin infection at the area of injection
* Coagulopathy
* History of allergy to local anaesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery | At 24 hours post surgery
  Comparing the quality of recovery 15 (QoR15) score at 24 hours between the study groups. QoR15: a minimum score of 0 (poor recovery) and a maximum score of 150 (excellent recovery)

SECONDARY OUTCOMES:
Area under the curve for pain at rest and movement (deep breathing) | Over the first 24 hours after surgery
  Comparing the area under the curve (AUC) of postoperative pain numerical rating score (NRS, 0-10) at rest and deep breathing (pain burden).
Number of hypoesthetic and anaesthetic dermatomes | At 15 and 30 minutes after block completion
  Number of anaesthetic and hypoesthetic dermatomes on the ventral and dorsal aspect of the thorax
Rescue fentanyl and phenylephrine administration | Intraoperative
  Total rescue fentanyl and phenylephrine administration
Postoperative morphine, tramadol and ondansetron consumption | At 24 and 48 hour post sugery
  Total postoperative morphine, tramadol and ondansetron consumption

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, FRCA, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Anaesthesia, Pain and Perioperative Medicine, Prince of Wales Hospital, Shatin, New Territories, Hong Kong